CLINICAL TRIAL: NCT03519282
Title: Clinical Evaluation of Biofinity Multifocal Toric Contact Lenses
Brief Title: Clinical Evaluation of Investigational Multifocal Toric Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CV-18-11
Record Dates: First submitted 2018-04-26; First posted 2018-05-08 (Actual); Results first posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Presbyopia; Astigmatism
MeSH Terms: conditions — Presbyopia; Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test Multifocal Toric Lens (Experimental): comfilcon A multifocal toric lens
  Interventions: Device: comfilcon A multifocal toric lens; Device: omafilcon A Multifocal Toric Lens
- omafilcon A Multifocal Toric Lens (Active Comparator): Control multifocal toric lens
  Interventions: Device: comfilcon A multifocal toric lens; Device: omafilcon A Multifocal Toric Lens

INTERVENTIONS:
Device: comfilcon A multifocal toric lens — contact lens
  Other Names: Test Multifocal Toric Lens; Biofinity multifocal toric lens
Device: omafilcon A Multifocal Toric Lens — contact lens
  Other Names: Proclear multifocal toric lens; Control multifocal toric lens

SUMMARY:
This non-dispensing study is to evaluate the clinical performance of a test multifocal toric silicone hydrogel contact lens compared to a marketed multifocal toric contact lens (control).

DETAILED DESCRIPTION:
This non-dispensing study is to evaluate the clinical performance of a test multifocal toric silicone hydrogel contact lens compared to a marketed multifocal toric contact lens (control).

ELIGIBILITY:
Inclusion Criteria:

* Has had a self-reported oculo-visual examination in the last two years.
* Is aged 40-75 years, inclusive and has full legal capacity to volunteer.
* Has read and understood the participant information sheet.
* Is willing and able to follow instructions and maintain the appointment schedule.
* Is able to participate in Parts A and B related to this work.
* Has a contact lens spherical prescription between +10.00 to -10.00D (inclusive).
* Has an Add component to their spectacle refraction (between +0.75 and +2.50DS).
* Has astigmatism between -0.75 and -5.75DC (based on the vertexed ocular refraction in each eye.
* Can be satisfactorily fitted with the study lenses.
* Is correctable to a visual acuity of 20/40 (0.30 logMAR) or better (in each eye) with their habitual vision correction or 20/25 (0.10 logMAR) best-corrected.
* They have successfully worn soft contact lenses in the last six months
* Has clear corneas and no active ocular disease.
* Has not worn lenses for at least 12 hours before the examination.
* Has an up-to-date pair of spectacles.

Exclusion Criteria:

* Has never worn contact lenses before.
* Has any systemic disease affecting ocular health.
* Is using any systemic or topical medications that will affect ocular health.
* Has any ocular pathology or severe insufficiency of lacrimal secretion (moderate to severe dry eyes) that would, in the opinion of the investigator, affect the wearing of contact lenses.
* Has persistent, clinically significant corneal or conjunctival staining using sodium fluorescein dye that would, in the opinion of the investigator, be problematic for their participation in the study.
* Has any clinically significant lid or conjunctival abnormalities, active neovascularization or any central corneal scars.
* Is aphakic.
* Has undergone corneal refractive surgery.
* Has a history of anaphylaxis or severe allergic reaction.
* Has diabetes or an infectious or immunosuppressive disease which could contraindicate contact lens wear or pose a risk to the investigator.
* They are pregnant or breast-feeding.
* Is participating in any other type of eye-related clinical or research study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2018-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Morgan, BSc, PhD, MCOptom, Principal Investigator — Eurolens Research
Locations (1):
- Eurolens Research, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three subjects did not meet the inclusion criteria. Ten (10) subjects completed all visits and their data were included in the analysis.
Groups:
- Test Multifocal Toric Lens Then Control Multifocal Toric: Subjects were randomized to wear the test multifocal toric lens then control multifocal toric lens during this crossover study.
  comfilcon A multifocal toric lens: contact lens
- Control Multifocal Toric Lens Then Test Multifocal Toric: Subjects were randomized to wear the control multifocal toric lens then test multifocal toric lens during this crossover study.
  omafilcon A Multifocal Toric Lens: contact lens
Period: First Intervention
Arm/Group | Test Multifocal Toric Lens Then Control Multifocal Toric | Control Multifocal Toric Lens Then Test Multifocal Toric
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Test Multifocal Toric Lens Then Control Multifocal Toric | Control Multifocal Toric Lens Then Test Multifocal Toric
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Comfilcon A and Omafilcon A Multifocal Toric Lenses: Subjects were randomized to wear the comfilcon A multifocal toric (test) or omafilcon A multifocal toric (control) lens, either as first or second lens during this cross over study.
Arm/Group | Comfilcon A and Omafilcon A Multifocal Toric Lenses
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 10

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Visual Acuity (measured in LogMAR)
Time Frame: Up to 2 hours
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Test Multifocal Toric Lens: Subjects were randomized to wear the comfilcon A multifocal toric lens during this crossover study.
  comfilcon A multifocal toric lens: contact lens
- Control Multifocal Toric Lens: Subjects were randomized to wear the omafilcon A Multifocal Toric Lens during this crossover study.
  omafilcon A Multifocal Toric Lens: contact lens
Arm/Group | Test Multifocal Toric Lens | Control Multifocal Toric Lens
Number analyzed (Participants) | 10 | 10
logMAR
  Distance: Binocular | -0.08 (0.05) | -0.06 (0.10)
  Distance: Monocular (dominate eye) | 0.00 (0.09) | -0.01 (0.06)
  Distant: Monocular (non-dominate eye) | 0.02 (0.09) | 0.01 (0.10)
  Near: Binocular | 0.10 (0.12) | 0.06 (0.12)
  Near: Monocular (dominate eye) | 0.15 (0.17) | 0.16 (0.17)
  Near: Monocular (non-dominate eye) | 0.17 (0.15) | 0.12 (0.14)

2. Secondary Outcome: Assessment of Visual Performance: Distance Navigation Tasks for Vision Quality and Clarity
Description: Subjective assessment of visual performance for distance navigation tasks for vision quality and clarity was assessed on a scale 0-100, 0=poor, 100=excellent.
Time Frame: Up to 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Multifocal Toric Lens | Control Multifocal Toric Lens
Number analyzed (Participants) | 10 | 10
units on a scale | 93 (9) | 87 (16)

3. Secondary Outcome: Assessment of Visual Performance: Intermediate Task for Vision Quality and Clarity
Description: Subjective assessment of visual performance for intermediate task for vision quality and clarity was assessed on a scale 0-100, 0=poor, 100=excellent.
Time Frame: Up to 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Multifocal Toric Lens | Control Multifocal Toric Lens
Number analyzed (Participants) | 10 | 10
units on a scale | 95 (9) | 95 (9)

4. Secondary Outcome: Assessment of Visual Performance: Near Task for Vision Quality and Clarity
Description: Subjective assessment of visual performance for near task for vision quality and clarity was assessed on a scale 0-100, 0=poor, 100=excellent.
Time Frame: Up to 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Multifocal Toric Lens | Control Multifocal Toric Lens
Number analyzed (Participants) | 10 | 10
units on a scale | 94 (8) | 90 (20)

ADVERSE EVENTS:
Time Frame: Up to 2 hours
Groups:
- Test Multifocal Toric Lens: Subjects were randomized to wear the comfilcon A multifocal toric lens, either as first or second lens during this crossover study.
  comfilcon A multifocal toric lens: contact lens
  omafilcon A Multifocal Toric Lens: contact lens
- Omafilcon A Multifocal Toric Lens: Subjects were randomized to wear the omafilcon A Multifocal Toric Lens, either as first or second lens during this crossover study.
  Control multifocal toric lens
  comfilcon A multifocal toric lens: contact lens
  omafilcon A Multifocal Toric Lens: contact lens
Arm/Group | Test Multifocal Toric Lens | Omafilcon A Multifocal Toric Lens
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT03519282/Prot_SAP_000.pdf